CLINICAL TRIAL: NCT05908786
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized Platform Study Evaluating The Efficacy and Safety of Neoadjuvant Immunotherapy Combinations in Patients With Surgically Resectable Hepatocellular Carcinoma (MORPHEUS-NEO HCC)
Brief Title: A Study Evaluating The Efficacy and Safety of Neoadjuvant Immunotherapy Combinations in Patients With Surgically Resectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO44457
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab; Tiragolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Atezo + Bev (Experimental): Participants in the atezolizumab plus bevacizumab (Atezo + Bev) arm will receive up to three cycles of treatment until surgery or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- Atezo + Bev +Tira (Experimental): Participants in the atezolizumab plus bevacizumab plus tiragolumab (Atezo + Bev +Tira) arm will receive up to three cycles of treatment until surgery or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Tiragolumab
- Tobe + Bev (Experimental): Participants in the Tobemstomig + Bev arm will receive up to three cycles of treatment until surgery or unacceptable toxicity, whichever occurs first.
  Enrollment is closed.
  Interventions: Drug: Bevacizumab; Drug: Tobemstomig

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a dose of 1200 mg by IV infusion on Day 1.
  Other Names: Tecentriq
  Arms: Atezo + Bev; Atezo + Bev +Tira
Drug: Bevacizumab — Bevacizumab will be administered at a dose of 15 mg/kg by IV infusion on Day 1.
  Other Names: Avastin
Drug: Tiragolumab — Tiragolumab will be administered at a dose of 600 mg by IV infusion on Day 1.
  Arms: Atezo + Bev +Tira
Drug: Tobemstomig — Tobemstomig will be administered at a dose of 600 mg by IV infusion on Day 1
  Other Names: RO7247669
  Arms: Tobe + Bev

SUMMARY:
This is a Phase Ib/II, open-label, multicenter, randomized platform study to evaluate neoadjuvant immunotherapy combinations in participants with resectable HCC. The study is designed with the flexibility to open new treatment arms as new agents become available, close existing treatment arms that demonstrate minimal clinical activity or unacceptable toxicity, or modify the participant population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HCC confirmed either histologically or clinically according to AASLD criteria for patients with cirrhosis. For participants without cirrhosis, histological confirmation is mandatory.
* HCC that is amenable to R0 surgical resection with curative intent in the opinion of the surgeons and oncologists or hepatologists involved in the care of the participant. Patients presenting with resectable HCC within or beyond Milan criteria (without extrahepatic spread or macrovascular invasion) are eligible.
* Measurable disease (at least one target lesion) according to RECIST v1.1 as determined by the investigator
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 within 7 days prior to randomization
* Child-Pugh Class A within 7 days prior to randomization
* Negative HIV test at screening
* No prior locoregional or systemic treatment for HCC
* Adequate hematologic and end-organ function
* Documented virology status of hepatitis
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating sperm

General Exclusion Criteria:

* Presence of extrahepatic disease or macrovascular invasion
* Known fibrolamellar HCC, sarcomatoid HCC, mixed cholangiocarcinoma and HCC, or other rare variants of HCC
* History of hepatic encephalopathy if clinically significant within one year prior to initiation of study treatment
* Moderate or severe ascites
* Active co-infection with HBV and HCV
* Known active co-infection with HBV and hepatitis D viral infection
* Prior treatment with CD137 agonists or immune checkpoint inhibitors, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or that are at high risk for bleeding
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment
* Inadequately controlled hypertension
* History of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease within 6 months prior to initiation of study treatment
* History of hemoptysis within 1 month prior to initiation of study treatment
* Evidence of bleeding diathesis or significant coagulopathy
* Current or recent (<= 10 days prior to initiation of study treatment) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes
* History of abdominal or tracheoesophageal fistula, GI perforation or intra-abdominal abscesses within 6 months prior to initiation of study treatment
* History of intestinal obstruction and/or clinical sign or symptoms of GI obstruction
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
* Grade >= proteinuria
* Major surgical procedure, open biopsy, or significant traumatic injury, or abdominal surgery, interventions or traumatic injuries, or anticipation of need of major surgical procedure other than potentially curative liver resection
* Chronic daily treatment with a non-steroidal anti-inflammatory drug (NSAID)
* Serious infection requiring oral or IV antibiotics and/or hospitalization
* Active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Major Pathologic Response (MPR) Rate | At the time of surgery
  MPR rate is defined as the proportion of participants with =<10% residual viable tumor in the tumor bed at the time of surgery, as assessed by central pathological review.

SECONDARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | At the time of surgery
  pCR rate is defined as the proportion of participants with an absence of residual tumor at the time of surgery, as assessed by central pathological review.
Relapse-Free Survival (RFS) | Surgery to the first documented recurrence of disease (up to approximately 2 years)
  RFS is defined as the time from surgery to the first documented recurrence of disease (intrahepatic or extrahepatic) according to EASL and/or RECIST v1.1, or death from any cause.
Event-Free Survival (EFS) | Randomization up to approximately 3 years
  EFS is defined as the time from randomization to any of the following events (whichever occurs first): disease progression that precludes surgery, as assessed by the investigator according RECIST v1.1; local regional, or distant disease recurrence as measured by EASL and/or RECIST v1.1; or death from any cause.
Overall Survival (OS) | Randomization to death from any cause (up to approximately 3 years)
  OS is defined as the time from randomization to death from any cause.
OS Rate at 24 Months | Randomization up to 24 months
  OS rate at 24 months is defined as the proportion of participants who have not experience death from any cause at 24 months after randomization.
OS Rate at 36 Months | Randomization up to 36 months
  OS rate at 36 months is defined as the proportion of participants who have not experience death from any cause at 36 months after randomization.
Objective Response Rate (ORR) | Prior to surgery
  ORR is defined as the proportion of participants with a radiographic Complete Response (CR) or Partial Response (PR) prior to surgery, as determined by the investigator according to RECIST v1.1 and HCC mRECIST. Responses will be assessed and determined according to RECIST v1.1 and HCC mRECIST but are not required to be confirmed by subsequent imaging assessments.
Proportion of Participants Downstaged to Within Milan Criteria | Prior to surgery
  Proportion of participants downstaged to within Milan criteria (for participants beyond criteria at randomization). Within Milan criteria is defined as single tumor <= 5 cm or 2 - 3 nodules all <= 3 cm.
R0 Resection Rate | At the time of surgery
  R0 resection rate (proportion of resected participants obtaining an R0 resection). R0 resection is defined as a microscopically margin-negative resection, in which no tumor (gross or microscopic) remains in the primary tumor bed.
Percentage of Participants With Adverse Events | Up to approximately 3 years after first participant enrolled
Proportion of Participants With Delayed or Canceled Surgery Due to Treatment-Related Adverse Events | >28 days from surgical restaging visit, anticipated up to 56 days
  Proportion of participants with delayed or canceled surgery due to treatment-related adverse events (defined as > 28 days from surgical restaging visit).
Post-Operative Surgical Complication Rates According to The Clavien-Dindo Surgical Classification | Surgery to treatment completion/discontinuation (up to approximately 2 years)
  Post-operative surgical complication rates according to the Clavien-Dindo surgical classification. Clinically relevant complications are defined as Clavien-Dindo Grade >= IIIa.
Post-Operative Mortality | Within 90 days after surgery
  Post-operative mortality is defined as death within 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- United States (6):
  - University of Southern California (USC), Los Angeles, California
  - University of California Los Angeles (UCLA) - Cancer Care - Santa Monica, Santa Monica, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Barbara Ann Karmanos Cancer Institute - Karmanos Cancer Center - Main Campus, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - UT Southwestern Medical Center, Dallas, Texas
- Austria (3):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Wiener Gesundheitsverbund, Klinik Favoriten, Vienna
  - Department of Internal Medicine III AKH and Medical University of Vienna, Vienna
- France (4):
  - Centre Georges Francois Leclerc (CGFL), Dijon
  - Centre Eugene Marquis (CEM), Rennes
  - Assistance Publique-Hopitaux de Paris, Villejuif
  - Gustave Roussy, Villejuif
- Germany (3):
  - University Essen, Essen
  - Universitaets Klinikum Frankfurt - Zentrum der Inneren Medizin, Frankfurt
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
- Auckland District Health Board (ADHB), Auckland, New Zealand
- South Korea (3):
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinic de Barcelona (Hospital Clinic i Provincial), Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
- Taiwan (5):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Medical Foundation, Kaohsiung Chang Gung Memorial Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital (NTUH) - Cancer Research Center, Zhongzheng Dist.
- Imperial College London - Imperial Centre for Translational and Experimental Medicine (ICTEM), London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing